CLINICAL TRIAL: NCT04682730
Title: An Implementation Strategy for the Adoption of an Evidence-Based Guideline for Pit-and-Fissure Sealants: Using a Framework From Organizational Development
Brief Title: An Implementation Strategy for the Adoption of an Evidence-Based Guideline for Pit-and-Fissure Sealants
Acronym: DISGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Deborah Polk, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY20020201; U01DE027452 (NIH); 17-077-E (Other: NIDCR)
Record Dates: First submitted 2020-12-16; First posted 2020-12-24 (Actual); Results first posted 2023-03-15 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Pit-and-Fissure Sealants
Keywords: evidence-based clinical practice guideline; dental sealants; Deliberative Democracy; Deliberative Loop

STUDY DESIGN:
Intervention Model Description: Stepped wedge. In addition to the vanguard clinic, there will be five steps, each with three clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deliberative Loop (Experimental): 28-page Context-Setting Document; 2-page addendum to Context-Setting Document; 90 minute Deliberative session; 8-page post-session survey
  Interventions: Behavioral: Deliberative Loop

INTERVENTIONS:
Behavioral: Deliberative Loop — The investigators will give background information to the stakeholders before they engage in the Deliberative session.
  Stakeholders from a given clinic will come together for a Deliberative session (i.e., facilitated conversation), enabling them to hear the full range of perspectives held by their fellow colleagues and to share their own perspective regarding how best to implement the guideline in small-group discussions.
  Following the Deliberative session, each stakeholder will have the opportunity to record their opinions regarding possible implementation interventions. The investigators will share these opinions with the clinic's decision-makers to help guide their decision-making about which implementation interventions to deploy. If a stakeholder happens to be absent the day of their clinic's Deliberative session, they will still have the opportunity to complete the survey.

SUMMARY:
The purpose of this implementation science study is to determine whether Deliberative Loops are effective in increasing providers' adherence to the non-cavitated caries component of the American Dental Association's pit-and-fissure sealant evidence-based clinical practice guideline. The investigators use a stepped wedge design to randomly assign dental clinics to the Deliberative Loop intervention. In a Deliberative Loop, stakeholders receive background information, participate in a facilitated discussion, and share their views with leadership. The Deliberative Loop intervention is designed to help stakeholders form informed opinions; in this study, stakeholders will be forming informed opinions about the implementation interventions they think will increase their clinic's adherence to the guideline. The investigators hypothesize that compared with the pre-intervention period, following the intervention, providers will place or treatment plan sealants for significantly more occlusal non-cavitated carious lesions.

DETAILED DESCRIPTION:
The purpose of this implementation science study is to determine whether Deliberative Loops are effective in increasing providers' adherence to the non-cavitated caries component of the American Dental Association's pit-and-fissure sealant evidence-based clinical practice guideline. The investigators use a stepped wedge design to randomly assign dental clinics to the Deliberative Loop intervention. In a Deliberative Loop, stakeholders receive background information, participate in a facilitated discussion, and share their views with leadership. The Deliberative Loop intervention is designed to help stakeholders form informed opinions; in this study, stakeholders will be forming informed opinions about the implementation interventions they think will increase their clinic's adherence to the guideline. The investigators hypothesize that compared with the pre-intervention period, following the intervention, providers will place or treatment plan sealants for significantly more occlusal non-cavitated carious lesions (NCCL).

All persons employed by Kaiser Permanente Northwest or Permanente Dental Associates and who work in a Kaiser Permanente Northwest dental clinic at any level [e.g., part time, full time] will be eligible to participate in the study. This includes both service providers and front-of-the-house staff, approximately 1,200 employees.

This is a Stage III study.

Participating sites include the 16 general dental clinics of Kaiser Permanente Northwest. All clinics are located within the United States.

The estimated time from when the study opens to enrollment until completion of data collection is 16 months. It will take approximately one to two months for each individual participant to complete all study-related tasks, depending on how soon after the introductory session the Deliberative session can be scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Employed by Kaiser Permanente Northwest Dental or Permanente Dental Associates
* Work in a Kaiser Permanente Northwest dental clinic

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 896 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Polk, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD sharing plan includes sharing with other researchers all collected, deidentified IPD.
Supporting Information: Study Protocol
Time Frame: Data from this study may be requested from other researchers up to five years after the completion of the primary endpoint.
Access Criteria: The investigators will make available the study protocol, data dictionary, and de-identified dataset for analysis for researchers who contact the clinical site PI, Jeff Fellows, to facilitate and to provide context for any planned analysis.

REFERENCES:
- [Derived] Polk DE, Shah NH, Dawson T, Gruss I, Pihlstrom DJ, Kaplan CD, Guerrero EG, Fellows JL. Results from a cluster-randomized, stepped-wedge trial testing a deliberative engagement intervention to increase guideline adherence among U.S. oral health providers. Sci Rep. 2025 May 25;15(1):18180. doi: 10.1038/s41598-025-03236-9. PMID 40415002
- [Derived] Gruss I, Dawson T, Kaplan CD, Pihlstrom DJ, Fellows JL, Polk DE. Utilizing deliberative engagement for identifying implementation strategy priorities: lessons learned from an online deliberative forum with dental professionals. Implement Sci Commun. 2023 Sep 21;4(1):119. doi: 10.1186/s43058-023-00496-2. PMID 37735706
- [Derived] Gruss I, Dawson T, Kaplan CD, Pihlstrom DJ, Reich S, Fellows JL, Polk DE. Sharing voice during deliberative engagement to improve guideline adherence in dental clinics: findings from a qualitative evaluation of an online deliberative forum discussion. BMJ Open. 2023 Jul 5;13(7):e072727. doi: 10.1136/bmjopen-2023-072727. PMID 37407045
- [Derived] Polk D, Shah NH, Dawson T, Gruss I, Pihlstrom DJ, Kaplan CD, Guerrero EG, Fellows JL. Testing a Deliberative Democracy Engagement Intervention to Increase Guideline-Concordance Among Oral Health Providers: Results from the DISGO Cluster-Randomized, Stepped-Wedge Trial. Res Sq [Preprint]. 2023 May 4:rs.3.rs-2757518. doi: 10.21203/rs.3.rs-2757518/v1. PMID 37205489
- [Derived] Polk DE, Guerrero EG, Gruss I, Shah NH, Yosuf NM, Dawson T, Kaplan CD, Pihlstrom DJ, Fellows JL. Study protocol: A stepped-wedge, cluster-randomized trial of the effectiveness of a deliberative loop in identifying implementation strategies for the adoption of a dental sealant guideline in dental clinics. Implement Sci Commun. 2021 Aug 28;2(1):96. doi: 10.1186/s43058-021-00199-6. PMID 34454637

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All providers and staff at 16 intervention clinics at Kaiser Permanente (KP). Overall study - January 1, 2021 - December 31, 2021
Pre-assignment Details: This is a stepped wedge cluster randomized trial where dental clinics were randomized to the Deliberative Loop intervention. Clinics were randomized to one of five intervention periods. We randomized three clinics at a time. The goal was to have a six-week window in which to run the three clinics that are in a given step and then a week gap before the next step's six-week window starts.
Units Other Than Participants: Dental Clinic
Groups:
- Deliberative Loop (DL) Vanguard: January 1, 2021- March 22, 2021 (3 months) non intervention period
  March 23, 2021- December 31, 2021 (9 months) intervention period
- DL Cluster 1: January 1, 2021 - April 29, 2021 or May 12, 2021 (4 - 4.5 months) non-intervention
  April 30, 2021 or May 13, 2021 (7.5 - 8 months) intervention
- DL Cluster 2: January 1, 2021 - June 17 or June 21 or June 24, 2021 ( 5.5 - 6 months) non-intervention
  June 18 or June 22 or June 25, 2021 - December 31, 2021 (6 - 6.5 months) intervention
- DL Cluster 3: January 1, 2021 - July 1 or July 28 or August 8, 2021 ( 6 - 7.5 months) non-intervention
  July 2 or July 29 or August 9, 2021 - December 31, 2021 (4.5 - 6 months) intervention
- DL Cluster 4: January 1, 2021 - September 14 or October 7, 2021 ( 8.5 - 9 months) non-intervention
  September 15 or October 8, 2021 - December 31, 2021 (3 - 3.5 months) intervention
- DL Cluster 5: January 1, 2021 - September 23 or October 7 or October 28, 2021 ( 9 - 10 months) non intervention
  September 24 or October 8 or October 29, 2021 - December 31, 2021 ( 2 - 3 months) intervention
Period: Overall Study
Arm/Group | Deliberative Loop (DL) Vanguard | DL Cluster 1 | DL Cluster 2 | DL Cluster 3 | DL Cluster 4 | DL Cluster 5
Started | 47; 1 Dental Clinic | 166; 3 Dental Clinic | 190; 3 Dental Clinic | 164; 3 Dental Clinic | 131; 3 Dental Clinic | 198; 3 Dental Clinic
Intro Session | 48; 1 Dental Clinic | 80; 3 Dental Clinic | 83; 3 Dental Clinic | 68; 3 Dental Clinic | 60; 3 Dental Clinic | 58; 3 Dental Clinic
Deliberative Forum | 25; 1 Dental Clinic | 89; 3 Dental Clinic | 76; 3 Dental Clinic | 64; 3 Dental Clinic | 54; 3 Dental Clinic | 55; 3 Dental Clinic
Surveys Received | 8; 1 Dental Clinic | 70; 3 Dental Clinic | 55; 3 Dental Clinic | 42; 3 Dental Clinic | 48; 3 Dental Clinic | 30; 3 Dental Clinic
Completed | 8; 1 Dental Clinic | 70; 3 Dental Clinic | 55; 3 Dental Clinic | 42; 3 Dental Clinic | 48; 3 Dental Clinic | 30; 3 Dental Clinic (Out of 896 potential participants (providers and staff employed at 16 intervention clinics at KP) 253 completed all study components.)
Not Completed | 39; 0 Dental Clinic | 96; 0 Dental Clinic | 135; 0 Dental Clinic | 122; 0 Dental Clinic | 83; 0 Dental Clinic | 168; 0 Dental Clinic

BASELINE CHARACTERISTICS:
Population: The study participants were dental providers/staff & units analyzed were teeth of providers' patients. The 16 intervention clinic census at study start was 896 providers/staff. At study end, we received demographics of providers/staff at the 16 clinics & received data for 680 (data received in aggregate & we are not able to break it out by cluster.) Some staff are floaters & not assigned to 1 clinic. They rotate clinics & may have been counted several times, resulting in the census discrepancy.
Units Other Than Participants: Teeth
Groups:
- Study Participants - Deliberative Loop: 28-page Context-Setting Document; 2-page addendum to Context-Setting Document; 90 minute Deliberative session; 8-page post-session survey
  Deliberative Loop: The investigators will give background information to the stakeholders before they engage in the Deliberative session. Stakeholders from a given clinic will come together for a Deliberative session (i.e., facilitated conversation), enabling them to hear the full range of perspectives held by their fellow colleagues and to share their own perspective regarding how best to implement the guideline in small-group discussions.
  Following the Deliberative session, each stakeholder will have the opportunity to record their opinions regarding possible implementation interventions. The investigators will share these opinions with the clinic's decision-makers to help guide their decision-making about which implementation interventions to deploy. If a stakeholder happens to be absent the day of their clinic's Deliberative session, they will still have the opportunity to complete the survey.
Arm/Group | Study Participants - Deliberative Loop
Number analyzed (Participants) | 680
Number analyzed (Teeth) | 5983
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 671
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 549
  Male | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45
  Not Hispanic or Latino | 635
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13
  Asian | 97
  Native Hawaiian or Other Pacific Islander | 6
  Black or African American | 26
  White | 520
  More than one race | 8
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 680
Provider rate of placing or treatment planning sealants for occlusal NCCLs [Count of Units; unit: Teeth] | 137

OUTCOME MEASURES:

1. Primary Outcome: Change in Providers' Rates of Placing or Treatment Planning Sealants for Occlusal NCCLs
Description: The change in the providers' rates of placing or treatment planning sealants for occlusal NCCLs from before to after clinic stakeholders are exposed to the Deliberative Loop intervention
Time Frame: from one month before the first step to two months after the final step, 1 year.
Population: The study participants are dental providers/staff. However, our primary outcome measured the change in the dental providers' rates of placing or treatment planning sealants for occlusal NCCLs from before to after clinic stakeholders are exposed to the Deliberative Loop intervention. Therefore, the units analyzed were teeth of the providers' patients. The number of participant providers that apply to the 9600 teeth is not available.
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Groups:
- Deliberative Loop: 28-page Context-Setting Document; 2-page addendum to Context-Setting Document; 90 minute Deliberative session; 8-page post-session survey
  Deliberative Loop: The investigators will give background information to the stakeholders before they engage in the Deliberative session. Stakeholders from a given clinic will come together for a Deliberative session (i.e., facilitated conversation), enabling them to hear the full range of perspectives held by their fellow colleagues and to share their own perspective regarding how best to implement the guideline in small-group discussions.
  Following the Deliberative session, each stakeholder will have the opportunity to record their opinions regarding possible implementation interventions. The investigators will share these opinions with the clinic's decision-makers to help guide their decision-making about which implementation interventions to deploy. If a stakeholder happens to be absent the day of their clinic's Deliberative session, they will still have the opportunity to complete the survey.
Arm/Group | Deliberative Loop
Number analyzed (Participants) | NA
Number analyzed (Teeth) | 9600
Teeth
  Pre-intervention: number analyzed (Teeth) | 5983
  Pre-intervention | 137
  Post-intervention: number analyzed (Teeth) | 3617
  Post-intervention | 95
Statistical Analysis 1: Comparison: Deliberative Loop; Test type: Superiority; p = 0.18, Mixed Models Analysis; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.58 to 1.11], Standard Error of Mean 0.13

2. Secondary Outcome: Total Program Costs
Description: Program costs: Total intervention costs. Program cost analysis conducted for the Deliberative Loop (DL) intervention using an opportunity cost approach. Program costs were estimated for the DL intervention (Workbook development - including the guideline, EHR data analyses, initial practitioner survey, and evidence review - and printing; Online DL session facilitator training and delivery, and program tailoring; dental office staff time; costs for implemented strategies, if applicable; and allowed charges for dental sealant placements). All costs are reported in 2021 dollars. The study analysis period was Jan 1-Dec 31, 2021, and in 16 clinics during 2021.
Time Frame: from planning the survey to gather background information to two months after the final step; an average of 1 year
Population: KPNW Dental system
Measure: Number; unit: dollars
Units Other Than Participants: Dental System
Arm/Group | Deliberative Loop
Number analyzed (Participants) | NA
Number analyzed (Dental System) | 1
dollars | 125,521

3. Secondary Outcome: Cost Per Clinic
Description: Program costs: Cost per clinic
Time Frame: from planning the survey to gather background information to two months after the final step; an average of 1 year
Population: 16 dental clinics
Measure: Mean (95% Confidence Interval); unit: dollars per clinic
Units Other Than Participants: dental clinics
Arm/Group | Deliberative Loop
Number analyzed (Participants) | NA
Number analyzed (dental clinics) | 16
dollars per clinic | 7845 [6378 to 9312]
Statistical Analysis 1: Comparison: Deliberative Loop; Mean Total Program costs per clinic for the KPNW Dental system; Test type: Other — single intervention group across 16 clinics; mean total program costs in 2021 dollars = 7845, 95% CI 2-sided [6378 to 9312], Standard Deviation 2,753 — An opportunity cost approach was used. Costs estimated: Develop workbook- guideline, EHR data analyses, survey, evidence review- & print; facilitator training/delivery/program tailoring; staff time; implemented strategies; dental sealant placements

4. Secondary Outcome: Cost Per Member Per Month (PMPM)
Description: Total intervention costs per member per month. Program cost analysis conducted for the Deliberative Loop (DL) intervention using an opportunity cost approach. Program costs were estimated for the DL intervention (Workbook development - including the guideline, EHR data analyses, initial practitioner survey, and evidence review - and printing; Online DL session facilitator training and delivery, and program tailoring; dental office staff time; costs for implemented strategies, if applicable; and allowed charges for dental sealant placements). All costs are reported in 2021 dollars. The study analysis period was Jan 1-Dec 31, 2021, and in 16 clinics during 2021. There were 265,200 members age 6 years or more on January 1, 2021, or a total of 3,182,400 member months.
Time Frame: from planning the survey to gather background information to two months after the final step; an average of 1 year
Population: 265,200 members age 6 yrs or more on January 1, 2021 x 12 months.
Measure: Number; unit: dollars per member per month
Units Other Than Participants: Members/patients
Arm/Group | Deliberative Loop
Number analyzed (Participants) | NA
Number analyzed (Members/patients) | 3182400
dollars per member per month | 0.039

5. Secondary Outcome: Annualized Costs for Guideline Implementation Interventions
Description: Program costs: Annualized costs for guideline implementation interventions
Time Frame: from planning the survey to gather background information to two months after the final step; an average of 1 year
Population: KPNW Dental System. All costs reported are automatically annualized. Originally we thought the intervention would cross calendar years. Since the intervention took place entirely in 2021, it is automatically annualized.
Measure: Number; unit: dollars
Units Other Than Participants: dental system
Arm/Group | Deliberative Loop
Number analyzed (Participants) | NA
Number analyzed (dental system) | 1
dollars | 125,521

6. Secondary Outcome: NCCL Treatment Costs- Total Program Costs Per Sealant
Description: Total intervention costs per sealant. Program cost analysis conducted for the Deliberative Loop (DL) intervention using an opportunity cost approach. Program costs were estimated for the DL intervention (Workbook development - including the guideline, EHR data analyses, initial practitioner survey, and evidence review - and printing; Online DL session facilitator training and delivery, and program tailoring; dental office staff time; costs for implemented strategies, if applicable; and allowed charges for dental sealant placements). All costs are reported in 2021 dollars. The study analysis period was Jan 1-Dec 31, 2021, and in 16 clinics during 2021. There were 95 sealants placed during the intervention period at 16 clinics.
Time Frame: from planning the survey to gather background information to two months after the final step; an average of 1 year
Population: Within KPNW Dental system, teeth receiving a sealant.
Measure: Number; unit: dollars per sealant
Units Other Than Participants: teeth
Arm/Group | Deliberative Loop
Number analyzed (Participants) | NA
Number analyzed (teeth) | 95
dollars per sealant | 1321

7. Secondary Outcome: NCCL Treatment Costs- Total Program Costs Per Sealant Per Clinic
Description: Program costs: NCCL treatment costs- Total program costs per sealant per clinic
Time Frame: from planning the survey to gather background information to two months after the final step; an average of 1 year
Population: KPNW Dental System / 16 intervention clinics
Measure: Mean (95% Confidence Interval); unit: dollars per sealant per clinic
Units Other Than Participants: dental clinics
Arm/Group | Deliberative Loop
Number analyzed (Participants) | NA
Number analyzed (dental clinics) | 16
dollars per sealant per clinic | 1321 [845 to 3208]
Statistical Analysis 1: Comparison: Deliberative Loop; Mean Total Program costs per sealant per clinic for the KPNW Dental system; Test type: Other — single intervention group across 16 clinics; mean total costs/per clinic per sealant = 1321, 95% CI 2-sided [845 to 3208], Standard Deviation 1245 — Total cost per sealant calculated as quotient of total intervention costs ($125,521) & total sealants placed (95), is = to mean cost/sealant across each clinic ($7845/5.938)

8. Secondary Outcome: NCCL Treatment Costs- Per Sealant Per Member Per Month (PMPM)
Description: Total intervention costs per sealant per member per month. Program cost analysis conducted for the Deliberative Loop (DL) intervention using an opportunity cost approach. Program costs were estimated for the DL intervention (Workbook development - including the guideline, EHR data analyses, initial practitioner survey, and evidence review - and printing; Online DL session facilitator training and delivery, and program tailoring; dental office staff time; costs for implemented strategies, if applicable; and allowed charges for dental sealant placements). All costs are reported in 2021 dollars. The study analysis period was Jan 1-Dec 31, 2021, and in 16 clinics during 2021. There were 95 sealants placed during the intervention period at 16 clinics. There were 265,200 members age 6 years or more on January 1, 2021, or a total of 3,182,400 member months.
Time Frame: from planning the survey to gather background information to two months after the final step; an average of 1 year
Population: 265,200 members age 6 yrs or more on Jan1, 2021
Measure: Number; unit: dollars per sealant PMPM
Units Other Than Participants: Members/patients
Arm/Group | Deliberative Loop
Number analyzed (Participants) | NA
Number analyzed (Members/patients) | 265200
dollars per sealant PMPM | 0.0004

9. Secondary Outcome: Sealant Treatment Plan Resolution
Description: The count of occlusal NCCLs with a treatment plan for sealants that is sealed by the end of the post-intervention evaluation period.
Time Frame: when a clinic was exposed to the intervention (when they received their survey results) to December 31, 2021. (Vanguard- 9.34 months; Cluster 1- 7.84 months; Cluster 2- 6.39 months; Cluster 3- 5.30 months; Cluster 4- 3.33 months; Cluster 5- 2.75 months)
Population: Teeth with a treatment plan
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Deliberative Loop
Number analyzed (Participants) | NA
Number analyzed (Teeth) | 89
Teeth | 89
Statistical Analysis 1: Comparison: Deliberative Loop; Test type: Other — descriptive analysis; percentage = 100; 89/89 treatment plans completed by the end of the period

10. Secondary Outcome: Cost Effectiveness
Description: Estimated incremental cost-effectiveness ratios (ICERs) for clinics after exposure to the intervention. ICERs calculated for annualized total costs, costs per clinic, and costs PMPM.
Time Frame: from one month before the first step to two months after the final step, 1 year
Population: Cost-effectiveness analyses are not conducted for interventions that are found to be ineffective compared to controls. Therefore, measure could not be assessed due to the results of the primary outcome measure.
Arm/Group | Deliberative Loop
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Acceptability, Management - Deliberative Loop Process
Description: management's perceptions of the acceptability of the Deliberative Loop process measured on a 5-point Likert scale, 0=not at all acceptable to 4=completely acceptable
  These ratings were dependent upon having all other analyses completed.
Time Frame: A single assessment following completion of all data analyses, approximately 1.5 years after the data collection end date.
Population: PDA Dental Director for Evidence Based Practice - this is one person
Measure: Number; unit: score on a scale
Arm/Group | Deliberative Loop
Number analyzed (Participants) | 1
score on a scale | 1.5

12. Other Pre Specified Outcome: Acceptability, Stakeholders - Deliberative Loop Process
Description: Stakeholders' perceptions of the acceptability of the Deliberative Loop process, 1 question, 5-point Likert scale, 0=Strongly Disagree, 4=Strongly Agree
  A higher score means more acceptability.
  Note: UBT stands for unit-based team. It is a group of frontline employees, including managers, dental staff (assistants, hygienists), and dentists who work together. UBTs hold regular meetings as part of their standard work flow and collaborate with one another to improve member and patient care.
Time Frame: One survey was available for participants to complete immediately following the deliberative loop session and the survey stayed available for 1 week following the deliberative loop session.
Population: Participants in deliberative loop process and UBT process. Same participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deliberative Loop
Number analyzed (Participants) | 206
score on a scale
  Deliberative Loop | 1.9 (1.3)
  UBT: number analyzed (Participants) | 195
  UBT | 2.7 (1.0)

13. Other Pre Specified Outcome: Acceptability, Stakeholders - Context Setting Document
Description: Stakeholders' perceptions of the acceptability of the Context-Setting Document, 3 questions measured on a 5-point Likert scale, 0=Strongly disagree to 12=Strongly agree. Note - Each item is 0 to 4, and the total score ranges from 0 - 12.
  A higher score means more acceptability.
Time Frame: as for outcome 12
Population: Post deliberative loop session survey respondents.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deliberative Loop
Number analyzed (Participants) | 213
score on a scale | 6.4 (3.0)

14. Other Pre Specified Outcome: Helpfulness of Group Discussion
Description: Stakeholders' perceptions of helpfulness of group discussion measured on a 3 question, 5-point Likert scale, 0=Strongly disagree to 12=Strongly agree. Note - Each item is 0 to 4, and the total score ranges from 0 - 12.
  A higher score means more helpfulness.
  Note: UBT stands for unit-based team. It is a group of frontline employees, including managers, dental staff (assistants, hygienists), and dentists who work together. UBTs hold regular meetings as part of their standard work flow and collaborate with one another to improve member and patient care.
Time Frame: as for outcome 12
Population: Participants in both deliberative loop and UBT sessions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deliberative Loop
Number analyzed (Participants) | 217
score on a scale
  Deliberative loop helpfulness | 5.1 (3.0)
  UBT helpfulness: number analyzed (Participants) | 216
  UBT helpfulness | 8.3 (2.3)

15. Other Pre Specified Outcome: Promotive Voice
Description: Stakeholders' perceptions of ability to express new ideas or suggestions for improving the clinic, 5 questions, 5-point Likert scale. Note - Each item is 0 to 4, and the total score ranges from 0-20, 0=Strongly disagree to 20=Strongly agree.
  A higher score means more promotive voice.
  Note: UBT stands for unit-based team. It is a group of frontline employees, including managers, dental staff (assistants, hygienists), and dentists who work together. UBTs hold regular meetings as part of their standard work flow and collaborate with one another to improve member and patient care.
Time Frame: as for outcome 12
Population: Participants in both deliberative loop and UBT sessions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deliberative Loop
Number analyzed (Participants) | 217
score on a scale
  Deliberative Loop | 11.5 (5.4)
  UBT: number analyzed (Participants) | 204
  UBT | 15.4 (4.3)

16. Other Pre Specified Outcome: Prohibitive Voice
Description: Stakeholders' perceptions of ability to express concern about work practices that may be harmful to the clinic, 5 questions, 5-point Likert scale. Note - Each item is 0 to 4, and the total score ranges from 0-20, 0=Strongly disagree to 20=Strongly agree.
  A higher score means more prohibitive voice.
  Note: UBT stands for unit-based team. It is a group of frontline employees, including managers, dental staff (assistants, hygienists), and dentists who work together. UBTs hold regular meetings as part of their standard work flow and collaborate with one another to improve member and patient care.
Time Frame: as for outcome 12
Population: Participants in both deliberative loop and UBT sessions. Same participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deliberative Loop
Number analyzed (Participants) | 217
score on a scale
  Deliberative Loop | 10.7 (5.0)
  UBT: number analyzed (Participants) | 205
  UBT | 13.3 (4.5)

17. Other Pre Specified Outcome: Future Leadership Responsiveness
Description: Stakeholders' perceptions that suggestions will be taken into consideration by leadership, 1 item, 5-point Likert scale, 0=Strongly disagree to 4=Strongly agree
  A higher score means more leadership responsiveness.
Time Frame: as for outcome 12
Population: Participants in deliberative loop session who filled out the post-session survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deliberative Loop
Number analyzed (Participants) | 212
score on a scale | 2.4 (1.1)

18. Other Pre Specified Outcome: Past Leadership Responsiveness
Description: Stakeholders' perceptions that suggestions have been taken into consideration by leadership in the past, 2 questions, 5-point Likert scale. Note - Each item is 0 to 4, and the total score ranges from 0-8, 0=Strongly disagree to 8=Strongly agree.
  A higher score means more stakeholder perception of leadership responsiveness.
Time Frame: as for outcome 12
Population: Participants in the deliberative loop session who filled out the post-session survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deliberative Loop
Number analyzed (Participants) | 218
score on a scale | 4.4 (2.2)

19. Other Pre Specified Outcome: Overall Voice
Description: Stakeholders' perceptions of voice, 1 question, 5-point Likert scale, 0=Strongly disagree to 4=Strongly agree
  A higher score means more overall voice.
  Note: UBT stands for unit-based team. It is a group of frontline employees, including managers, dental staff (assistants, hygienists), and dentists who work together. UBTs hold regular meetings as part of their standard work flow and collaborate with one another to improve member and patient care.
Time Frame: as for outcome 12
Population: Participants in both deliberative loop and UBT sessions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deliberative Loop
Number analyzed (Participants) | 206
score on a scale
  Deliberative Loop Session | 1.9 (1.3)
  UBT Session: number analyzed (Participants) | 195
  UBT Session | 2.7 (1.0)

20. Other Pre Specified Outcome: Perceptions of Discussion
Description: Stakeholders' perceptions about the discussion, 2 questions, 5-point Likert scale. Note - Each item is 0 to 4, and the total score ranges from 0 - 8, 0=Strongly disagree to 8=Strongly agree.
  A higher score means more consideration of important issues and points of view.
  Note: UBT stands for unit-based team. It is a group of frontline employees, including managers, dental staff (assistants, hygienists), and dentists who work together. UBTs hold regular meetings as part of their standard work flow and collaborate with one another to improve member and patient care.
Time Frame: as for outcome 12
Population: Participants in both deliberative loop and UBT sessions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deliberative Loop
Number analyzed (Participants) | 203
score on a scale
  Deliberative Loop Session | 4.1 (2.2)
  UBT Session: number analyzed (Participants) | 197
  UBT Session | 5.6 (1.9)

21. Other Pre Specified Outcome: List of Implementation Strategies Endorsed by Stakeholders
Description: Stakeholders' informed opinion about what implementation strategies their clinic should adopt for each barrier
Time Frame: as for outcome 12
Reporting Status: Not Posted

22. Other Pre Specified Outcome: List of Barriers Perceived by Stakeholders
Description: Stakeholders' informed opinion about barriers they perceive in their clinic
Time Frame: One survey was available for participants to complete immediately following the DL session and the survey stayed available for 1 week following the session.
Reporting Status: Not Posted

23. Other Pre Specified Outcome: List of Implementation Strategies Adopted by the Clinics, Quantitative
Description: List of implementation strategies. Clinic staff can select strategies on the list that their clinic has adopted to document progress of the implementation process
Time Frame: 3 months after receiving the clinic summary report
Reporting Status: Not Posted

24. Other Pre Specified Outcome: List of Implementation Strategies Adopted by the Clinics, Qualitative
Description: qualitative interviews of clinic staff, using the quantitative forms as the basis for the interview
Time Frame: 3 months after receiving the clinic summary report
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year in which AE and SAE data could have been collected.
Description: As participants were dental providers/staff and the ones exposed to the intervention, collection of AE was not applicable.
Arm/Group | Deliberative Loop
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT04682730/Prot_SAP_000.pdf